CLINICAL TRIAL: NCT00567736
Title: Prospective Randomized Controlled Multicentre Trial for Patients With Chronic Low Back Pain Comparing Disci/Rhus Toxicodendron Comp.®, Placebo and Waiting List Group
Brief Title: Efficacy of Disci/Rhus Toxicodendron Comp.®, in Patients With Chronic Low Back Pain
Acronym: DISCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: WALA Heilmittel GmbH (Other)
Responsible Party: Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center Berlin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DISCI-07; EudraCT-Nr. 2006-006390-24
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; complementary therapies
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Disci/Rhus toxicodendron comp.®
  Interventions: Drug: Disci/Rhus toxicodendron comp.®
- 2 (Placebo Comparator): placebo solution
  Interventions: Drug: placebo solution
- 3 (No Intervention): waiting list group

INTERVENTIONS:
Drug: Disci/Rhus toxicodendron comp.® — s.c. application 10 ml (1 ampul) in 5 to 10 parts on different back pain sites verum group 12 treatments: 8 in the first 4 weeks and 4 in the next 4 weeks
  Arms: 1
Drug: placebo solution — s.c. application 10 ml (1 ampul) in 5 to 10 parts on different back pain sites 12 treatments: 8 in the first 4 weeks and 4 in the next 4 weeks
  Arms: 2

SUMMARY:
The aim of the study is to evaluate the efficacy of Disci/Rhus toxicodendron. comp.® in patients with chronic low back pain compared to waiting list group, or placebo.

DETAILED DESCRIPTION:
Chronic low back pain is a significant health problem in industrialized countries. Use of complementary medicine is increasing in patients with low back pain. Until now there is no evidence for the efficacy of Disci/Rhus toxicodendron. comp.® in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 30 to 75 years
* Willingness of following the study protocol
* Clinical diagnosis of chronic low back pain
* Low back pain since at least 3 months
* Average pain intensity of at least 40 mm on VAS (0-100 mm) in the last 7 days
* In the last 4 weeks only oral NSAD and muscle relaxation treatment
* Effective oral contraception in woman
* Informed consent

Exclusion Criteria:

* Previous treatment with DISCI comp.
* Treatment with other than NSAID
* Routine use of pain drugs for other diseases
* Protrusio or prolapse of one or more intervertebral discs with neurological symptoms
* Previous spine surgery
* (Suspicious) infectious spondylopathy
* Low back pain because of malignant or infectious disease
* Other causes of back pain symptoms (e.g. M. Bechterev, M. Reiter)
* Congenital deformity of spine (without minor lordosis or kyphosis or scoliosis
* (Suspicious) osteoporosis with compression fracture
* (Suspicious) spinal stenosis
* Spondylolysis or spondylolisthesis
* Physiotherapy in the last four weeks or planed during trial
* Begin of a new treatment for low back pain
* Complementary treatment in the last four weeks or planed during trial
* Patients who are not able to cooperate in a sufficient way
* Patients with alcohol or substance abuse
* Participation in another clinical trial
* Severe chronical or acute disease which does not allow study participation
* Patients with bleeding disorders or oral anticoagulation treatment
* Pregnancy and breast feeding
* Patients with application for pension
* Patients involved in planning or coordination of the study
* Hypersensitivity against drug components

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (0-100 mm) low back pain | once after 8 weeks

SECONDARY OUTCOMES:
Back function (back function scale FFbHR) | once at week 8 and 26
visual analogue scale (0-100 mm) low back pain | once after week 26
days with medication | week 4 to 8
quality of life (SF-36) | once at week 8 and 26
pain disability scale (PDI) | once at week 8 and 26
emotional pain scale (SES) | once at week 8 and 26
influence of patient expectancy | once at week 8 and 26
influence of physician expectancy | once at week 8 and 26
Responder rate 36% VAS pain intensity | once at week 8 and 26
numbers of days with absence from work | between week 4 and 8
days with physician visits because of low back pain | between week 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- o Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany

REFERENCES:
- [Result] Pach D, Brinkhaus B, Roll S, Wegscheider K, Icke K, Willich SN, Witt CM. Efficacy of injections with Disci/Rhus toxicodendron compositum for chronic low back pain--a randomized placebo-controlled trial. PLoS One. 2011;6(11):e26166. doi: 10.1371/journal.pone.0026166. Epub 2011 Nov 8. PMID 22087222